CLINICAL TRIAL: NCT02197403
Title: Comparative Study on Development of Paradoxical Excitement Response During Sedation Using Dexmedetomidine or Propofol in Hazardous Alcohol Drinkers
Brief Title: Paradoxical Excitement Response During Sedation Between Dexmedetomidine and Propofol in Hazardous Alcohol Drinker
Acronym: DEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-il Choi, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: an00543
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia, Spinal; Sedation, Conscious; Dexmedetomidine; Alcohol Drinking; Anesthesia, Epidural; Propofol
Keywords: Dexmedetomidine; Sedation; Paradoxical excitement response; Alcohol drinkers
MeSH Terms: conditions — Alcohol Drinking | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- alcohol drinker & dexmedetomidine (Experimental): dexmedetomidine, 200mcg in 50mL of normal saline 0.75mcg/Kg bolus injection in 10 minutes 0.1~1.0mcg/Kg infusion during surgery
  Interventions: Drug: Dexmedetomidine
- alcohol drinker & propofol (Active Comparator): Propofol (2% fresofol) 25~75mcg/kg/min continuous infusion
  Interventions: Drug: Propofol
- Non-alcohol drinker & dexmedetomidine (Active Comparator): dexmedetomidine, 200mcg in 50mL of normal saline 0.75mcg/Kg bolus injection in 10 minutes 0.1~1.0mcg/Kg infusion during surgery
  Interventions: Drug: Dexmedetomidine
- Non-alcohol drinker & propofol (Active Comparator): Propofol (2% fresofol) 25~75mcg/kg/min continuous infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — 200mcg in 50mL of normal saline 0.75mcg/Kg bolus injection in 10 minutes 0.1~1.0mcg/Kg infusion
  Other Names: Precedex
  Arms: Non-alcohol drinker & dexmedetomidine; alcohol drinker & dexmedetomidine
Drug: Propofol — 25~75mcg/kg/min continuous infusion
  Other Names: Fresofol
  Arms: Non-alcohol drinker & propofol; alcohol drinker & propofol

SUMMARY:
1. Adequate sedation with classical sedative agents, propofol
2. Sedation with propofol may induce paradoxical excitement response in heavy alcohol drinkers
3. Dexmedetomidine, α2 receptor agonist, may provide adequate sedation in heavy alcohol drinkers

DETAILED DESCRIPTION:
1. Adequate sedation during surgery provide anxiolysis and comfort to patient. Insufficient sedation can't provide comfort to patient during surgery, otherwise excessive sedation can cause variable complications like respiratory depression or delayed awakening.
2. Dexmedetomidine is a centrally acting α2 receptor agonist that is increasingly being used as a sedative for MAC and intensive care with mechanical ventilated patients because of its analgesic properties, "cooperative sedation," and lack of respiratory depression.
3. Because of the different site of action between dexmedetomidine and propofol, we assumed that paradoxical excitement responses which appeared in heavy alcohol drinkers in midazolam or propofol-induced sedation might be less observed in dexmedetomidine-induced sedation.

ELIGIBILITY:
Inclusion Criteria:

* 19~65 yr-old patients who is scheduled to undergo knee surgery with regional anesthesia

Exclusion Criteria:

* History of taking anxiolytics, hypnotics, antiepileptic drugs
* Abnormal liver function test (eg: Liver cirrhosis, elevated liver enzymes)
* History of allergic reaction with dexmedetomidine or propofol
* Contraindication with regional anesthesia
* American society of anesthesiologist Physical status III or IV

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-12; Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Paradoxical excitement response | Every 5 minutes up to 120minutes after drug infusion
  Paradoxical excitement responses (verbal/movement) 0, none : no excitement response
  1. mild : increased talkativeness, irrational talking / brief spontaneous movement with position remaining
  2. moderate : restlessness, loss of cooperation, spontaneous movements requiring repositioning with no need of restraint
  3. severe : agitation and spontaneous movements with a need to restrain the patient

SECONDARY OUTCOMES:
OAA/S | Every 5minutes up to 120minutes after drug infusion
  Observer''s Assessment of Alertness/Sedation Scale (OAA/S)
  1. :Does not respond to mild prodding or shaking
  2. :Responds only after mild prodding or shaking
  3. :Responds only after name is spoken loudly and/or repeatedly
  4. :Lethargic response to name spoken in normal tone
  5. :Responds readily to name spoken in normal tone
  Goal to sedation : 3
Vital signs | During operation
  Check blood pressure, heart rate, oxygen saturation, bispectral index

CONTACTS AND LOCATIONS:
Overall Officials: Hyunjung Lee, MD, Master, Principal Investigator — Chonnam National University Hospital; Jeongil Choi, MD, PhD, Study Director — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanamdo, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jeong S, Lee HG, Kim WM, Jeong CW, Lee SH, Yoon MH, Choi JI. Increase of paradoxical excitement response during propofol-induced sedation in hazardous and harmful alcohol drinkers. Br J Anaesth. 2011 Dec;107(6):930-3. doi: 10.1093/bja/aer275. Epub 2011 Sep 7. PMID 21903640
- [Result] Adams R, Brown GT, Davidson M, Fisher E, Mathisen J, Thomson G, Webster NR. Efficacy of dexmedetomidine compared with midazolam for sedation in adult intensive care patients: a systematic review. Br J Anaesth. 2013 Nov;111(5):703-10. doi: 10.1093/bja/aet194. Epub 2013 Jun 7. PMID 23748199
- [Result] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955
- [Result] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256